CLINICAL TRIAL: NCT06449482
Title: An Exploratory Clinical Study of Selinexor Combined With Venetoclax and Azactidine in the Treatment of Acute Myeloid Leukemia Patients Who Are Not Eligible for Intense Chemotherapy Regimen at Initial Treatment
Brief Title: Selinexor、Venetoclax and Azactidine in the Treatment of ND AML Patients Who Are Not Eligible for Intense Chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The number of participants in the study did not meet expectations
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022053
Record Dates: First submitted 2023-06-13; First posted 2024-06-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; venetoclax; Azacitidine

STUDY DESIGN:
Intervention Model Description: selinexor venetoclax and azacitidine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- selinexor venetoclax Azacitidine (Experimental): In the dose-increasing stage, the subject induction therapy was designed using a 3+3 design. selinexor 60mg QW, 40mg BIW, or 60mg BIW, in combination with venetoclax 100mg d1 200mg d2 400mg d3-28, orally once a day, and azacitidine 75mg/m2, d1-7, subcutaneously. The medication regimen was repeated every 28 days. In this case, RP2D is determined based on MTD, safety, and all other data.
  During this study period, there were a total of 4 courses. The treatment cycle of the subjects will include 2 cycles of induction therapy and up to 2 cycles of consolidation therapy.
  Interventions: Drug: Selinexor; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Selinexor — three dosage groups were set up, selinexor 60mg QW, 40mg BIW, or 60mg BIW
  Other Names: XPO1-i
Drug: Venetoclax — cycle 1 100mg d1 200mg d2 400mg d3-28 cycle 2-4 400mg d1-d28
  Other Names: BCL-2i
Drug: Azacitidine — 75mg/m2 d1-d7 28d/cycle 4 cycles

SUMMARY:
This study is a single arm open exploratory clinical trial to evaluate the efficacy and safety of selinexor combined with venetoclax and azacitidine. This study will be divided into two stages: dose increasing stage and dose expanding stage. In the dose-increasing stage, the study induction therapy was designed using a 3+3 design. The induction therapy and consolidation therapy of the subjects will be administered at RP2D doses.

During this study period, there were a total of 4 cycles. The treatment cycle of the subjects will include 2 cycles of induction therapy and up to 2 cycles of consolidation therapy.

In addition, if the subject does not achieve remission (CR/Cr or PR) after 2 cycles of consolidation treatment (at the end of the 4th course), the study will be terminated by the subject, and the clinical doctor will choose the subsequent treatment for the subject based on clinical experience.

DETAILED DESCRIPTION:
This study is a single arm open exploratory clinical trial to evaluate the efficacy and safety of selinexor combined with venetoclax and azacitidine. This study will be divided into two stages: dose increasing stage and dose expanding stage. In the dose-increasing stage, the study induction therapy was designed using a 3+3 design. In this stage, three dosage groups were set up, namely selinexor 60mg QW, 40mg BIW, or 60mg BIW, in combination with venetoclax 100mg d1 200mg d2 400mg d3-28, orally once a day, and azacitidine 75mg/m2, d1-7, subcutaneously. The regimen was repeated every 28 days. In this case, RP2D is determined based on MTD, safety, and all other data.

The methods of venetoclax and azacitidine remain unchanged during consolidation therapy. Before RP2D is determined, the dosage of selinexor is determined by the researchers based on individual subject tolerance. After RP2D is determined, the study enters the second stage of dose expansion. The induction therapy and consolidation therapy of the subjects will be administered at RP2D doses.

During this study period, there were a total of 4 cycles. The treatment cycle of the subjects will include 2 cycles of induction therapy and up to 2 cycles of consolidation therapy. In addition, if the subject does not achieve remission (CR/Cr or PR) after 2 cycles of consolidation treatment (at the end of the 4th course), the study will be terminated by the subject, and the clinical doctor will choose the subsequent treatment for the subject based on clinical experience.

The subjects will participate in the screening period, treatment period, and follow-up period. The screening period lasts for a maximum of 28 days before medication. The treatment period lasts from the first day of the first cycle to the end of the study treatment. The follow-up period starts after the end of treatment and lasts for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML patients diagnosed according to WHO standards who are not suitable for the standard induction treatment regimen of cytarabine combined with anthracycline drugs due to age or comorbidities.
2. Age ≥ 75 years old, ECOG score 0-2 points; The patient's age range is 18-75 years old, with an ECOG score of 0-3.
3. Liver function meets the following criteria: total bilirubin<3 × Upper limit of normal range (ULN) (<75 years old), total bilirubin<1.5 × ULN (≥ 75 years old), AST<3 × ULN and ALT<3 × ULN.
4. Renal function meets the following criteria: creatinine clearance rate ≥ 30 mL/min (Cockroft-Gault formula).
5. Expected survival time greater than 6 months

Exclusion Criteria:

1. patient who has received BCL2 inhibitors, demethylation drugs, chemotherapy, CAR-T therapy, or other experimental therapies.
2. History of myeloproliferative tumors (MPN).
3. Cytogenetic low risk, such as t (8; 21), inv (16), t (16; 16) or t (15; 17).
4. Acute promyelocytic leukemia.
5. AML central nervous system (CNS) involvement.
6. Pregnancy or lactation period.
7. I underwent major surgery within 4 weeks before the first study medication.
8. Subjects with unstable or active cardiovascular diseases who meet any of the following criteria:
9. Symptomatic myocardial ischemia;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
RP2D of selinexor in this study | 1 year
  from the first day to the last day of the cycle

SECONDARY OUTCOMES:
MRD negative rate | up to 16 weeks
  MRD negative rate at the end of 2 cycles and 4 cycles of induction therapy
Compound complete response rate | up to 16 weeks
  From first dose of treatment to first day response is documented by evaluation
The time to compound complete response | up to 16 weeks
  From first dose of treatment to first day response is documented by evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China